CLINICAL TRIAL: NCT05944393
Title: Erector Spine Plane (ESP) Block for Analgesia in Pediatric Scoliosis Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 673/22
Record Dates: First submitted 2023-02-19; First posted 2023-07-13 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Scoliosis; Regional Anesthesia; Pediatric Anesthesia; Orthopedic Disorder of Spine
Keywords: erector spine plane block; neuromonitoring; pain management; multimodal analgesia
MeSH Terms: conditions — Scoliosis; Agnosia | interventions — Ropivacaine; Saline Solution

STUDY DESIGN:
Intervention Model Description: after being informed about the study and potential risks. All patients giving written consent will be randomized in a double-blind manner into 2 groups each one containing 25 patients, ESP group (n =25 ): The patients will receive Erector Spine Plane Block (ESP Block) after induction of general anesthesia.
  Control group (n =25 ): The patients will receive a placebo block after induction of general anesthesia
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Subjects will be randomized to one of two groups with a computer-generated arm assignment. The sealed envelopes will be opened immediately prior to nerve block. One group will receive a ESP block and the other will receive a placebo block. The provider performing the block will not be blinded, however all other members of the care team, the patient, and the investigator collecting data will be blinded to the randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESB block (Experimental): Patients will receive preoperative ultrasound-guided bilateral single-injection ESP blocks at one or two levels before incision with 10 mL 0.2% ropivacaine per single injection. Using appropriate sterile precautions, under general anesthesia, an ultrasound (Mindrey TE9) equipped with either a linear 15-6 megahertz (MHz), or a curvilinear 5-2 MHz transducer (habitus-dependent) used to identify the erector spine, transverse process, and paravertebral space. A 22G 0,7x80 mm echogenic block needle (Stimuplex Ultra 360)) is inserted in-plane from the cranial to caudal direction until the needle tip contacts the transverse process. 1-3mL is injected to confirm the proper injection plane by visualizing the spread deep to the erector spinae muscles and superficial to the transverse process. Block is completed with 10mL of 0,2% Ropivacaine. The needle is withdrawn, and the needle entry site is wiped clean.
  Interventions: Drug: Ropivacaine 0.2% Injectable Solution
- Placebo block (Experimental): Patients will receive preoperative ultrasound-guided bilateral single-injection ESP blocks at one or two levels before incision with 10 mL 0,9% normal saline per single injection. Using appropriate sterile precautions, under general anesthesia, an ultrasound (Mindrey TE9) equipped with either a linear 15-6 megahertz (MHz), or a curvilinear 5-2 MHz transducer (habitus-dependent) used to identify the erector spine, transverse process, and paravertebral space. A 22G 0,7x80 mm echogenic block needle (Stimuplex Ultra 360)) is inserted in-plane from the cranial to caudal direction until the needle tip contacts the transverse process. 1-3mL is injected to confirm the proper injection plane by visualizing the spread deep to the erector spinae muscles and superficial to the transverse process. Block is completed with 10mL of 0,9% normal saline. The needle is withdrawn, and the needle entry site is wiped clean.
  Interventions: Drug: Normal saline 0.9% Injectable Solution

INTERVENTIONS:
Drug: Ropivacaine 0.2% Injectable Solution — Ultrasound-guided Erector Spine Plane block with 10 mL 0.5% ropivacaine
  Arms: ESB block
Drug: Normal saline 0.9% Injectable Solution — Ultrasound-guided Erector Spine Plane block with 10 mL 0.9% normal saline
  Arms: Placebo block

SUMMARY:
Postoperative pain after scoliosis correction surgery is severe and usually requires long-term intravenous opioid therapy. Local anesthetic options are limited and include intrathecal opioids and epidural analgesia. However, they are rarely used due to side effects and inconsistent efficacy. The investigators describe an opioid-sparing multimodal analgesia regimen with bilateral erector spinae plane blocks.

DETAILED DESCRIPTION:
Posterior spinal fusion for scoliosis correction is extremely painful and usually requires long-term, high-dose opioid use for adequate perioperative analgesia. Neuromonitoring, i.e., motor-evoked and somatosensory-evoked potentials (SSEPs), are the current gold standard for preventing neurological damage. Local anesthesia is essential to multimodal analgesia, but options are limited. Intrathecal or epidural opioid injections of local anesthetics have been reported but are rarely used due to logistical complexity, side effects, and inconsistent analgesic efficacy. The erector spinae plane (ESP) block was first described in 2016 for thoracic neuropathic pain. It is a new interfacial plane technique. Easy to perform on patients without spinal deformities. It was successfully used for surgery in adults. However, even with ultrasound guidance, identifying bone markers in scoliosis patients is challenging. The investigators will treat patients for scoliosis with single-shot bilateral ESP blocks. The investigators aim to provide effective perioperative pain control and achieve intraoperative hemodynamic stability without compromising neuromonitoring.

ELIGIBILITY:
Inclusion Criteria:

* Patients < 18 years old undergoing scoliosis surgery

Exclusion Criteria:

* refusal to participate
* > 18 yo
* Chronic opioid use
* localized infection

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-09-08 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
pain score | Within 30 minutes of emergence from anesthesia
  NRS (numerical rating scale) score (0- no pain to 10 worst pain)
pain score - 60 minutes | Within 60 minutes of emergence from anesthesia
  NRS (numerical rating scale) score (0- no pain to 10 worst pain)
pain score - 90 minutes | Within 90 minutes of emergence from anesthesia
  NRS (numerical rating scale) score (0- no pain to 10 worst pain)
pain score - 120 minutes | Within 120 minutes of emergence from anesthesia
  NRS (numerical rating scale) score (0- no pain to 10 worst pain)
pain score - 6 hours | Within 6 hours of emergence from anesthesia
  NRS (numerical rating scale) score (0- no pain to 10 worst pain)
pain score - 12 hours | Within 12 hours of emergence from anesthesia
  NRS (numerical rating scale) score (0- no pain to 10 worst pain)
pain score - 24 hours | Within 24 hours of emergence from anesthesia
  NRS (numerical rating scale) score (0- no pain to 10 worst pain)
pain score - 48 hours | Within 48 hours of emergence from anesthesia
  NRS (numerical rating scale) score (0- no pain to 10 worst pain)

SECONDARY OUTCOMES:
total opioid consumption within first 24 hours | Second day following the procedure
  Total morphine milligram equivalents required by patients in the post-anesthesia care unit, prior to discharge from the outpatient surgery center. Following emergence from anesthesia, pain will be assessed in regular intervals, with administration of IV and oral opioids according to numeric rating scale and clinical assessment. Opioid administration stops when patient numerical rating score is <4, when patient endorses manageable pain level, when side effects of opioids are intolerable, or for other concerning clinical conditions as determined by the anesthesiologist of record.
opioid consumption - 48 hours | Within 48 hours of emergence from anesthesia
  Total morphine milligram equivalents required by patients in the post-anesthesia care unit, prior to discharge from the outpatient surgery center. Following emergence from anesthesia, pain will be assessed in regular intervals, with administration of IV and oral opioids according to numeric rating scale and clinical assessment. Opioid administration stops when patient numerical rating score is <4, when patient endorses manageable pain level, when side effects of opioids are intolerable, or for other concerning clinical conditions as determined by the anesthesiologist of record.
Nausea and Vomiting | Beginning with emergence from anesthesia and ending with discharge from the post-anesthesia care unit (0-48 hours postoperativly)
  This is a yes/no binary outcome measure defined by administration of any antiemetic drug in the post-anesthesia care unit.
NLR -12 hours | 12 hours postoperatively
  neutrophil/limphocyte ratio
PLR -12 hours | 12 hours postoperatively
  platelet/limphocyte ratio
NLR - 24 hours | 12 hours postoperatively
  neutrophil/limphocyte ratio
PLR - 24 hours | 12 hours postoperatively
  platelet/limphocyte ratio

CONTACTS AND LOCATIONS:
Overall Officials: Małgorzata Domagalska, PhD, Principal Investigator — Department of Palliative Medicine, University of Medical Sciences; Tomasz Kotwicki, Profesor, Study Chair — Department of Spine Diseases and Pediatric Orthopedics, University of Medical Sciences
Locations (1):
- Department of Spine Diseases and Pediatric Orthopedics, University of Medical Sciences, Poznań, Poland, Poznan, Wielkopolska, Poland

IPD SHARING:
Plan to Share IPD: Yes
The data presented in this study are available on request from the corresponding author.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available after completing the study- December 2024
Access Criteria: The data presented in this study are available on request from the corresponding author.